CLINICAL TRIAL: NCT00083564
Title: A Randomized Multicenter Study to Compare the Safety and Efficacy of 166Ho-DOTMP Plus Melphalan to Melphalan Alone as Conditioning for Autologous Peripheral Blood Stem Cell Transplant in Subjects With Primary Refractory Multiple Myeloma
Brief Title: Study Comparing STR (Skeletal Targeted Radiotherapy) Plus Melphalan to Melphalan Alone, With Stem Cell Transplant in Multiple Myeloma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: For business reasons
Sponsor: Poniard Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STR 0303
Record Dates: First submitted 2004-05-25; First posted 2004-05-28 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Primary refractory multiple myeloma; STR; Skeletal Targeted Radiotherapy; Holmium-166; 166-Ho-DOTMP
MeSH Terms: conditions — Multiple Myeloma | interventions — holmium-1,4,7,10-tetraazacyclododecane-N,N',N'',N'''-tetrakis(methylenephosphonic acid)

INTERVENTIONS:
Drug: STR(TM) (Skeletal Targeted Radiotherapy, Holmium-166-DOTMP)

SUMMARY:
STR (Skeletal Targeted Radiotherapy, 166Ho-DOTMP) is an investigational radiopharmaceutical that delivers radiation directly to cancer cells in the bone and bone marrow. Conventional methods of delivering radiation therapy, such as total body irradiation, expose non-target tissues to radiation and cause serious side effects. In contrast, STR's targeted approach to delivering radiotherapy concentrates the radiation where it is needed, and minimizes exposure of normal tissues.

STR is composed of a bone-targeting molecule, DOTMP, in a stable complex with the radionuclide holmium-166. When injected into a patient's bloodstream, STR rapidly binds to bone mineral, delivering a brief, intense dose of radiation to destroy cancer cells in the bone and marrow. The high-energy and long path-length of holmium-166 beta particles provide optimal penetration and uniform irradiation of disease sites in the marrow and bone. STR that does not bind to bone is rapidly eliminated through the urinary tract. STR treatment is followed by autologous stem cell transplantation. The short half-life of holmium-166 allows treatment on an out-patient basis, and minimizes the time required between STR administration and transplantation.

The phase III study of STR is a multi-center, randomized, controlled study, designed to evaluate the safety and efficacy of STR in patients with primary refractory multiple myeloma. These are patients who have failed to achieve at least a partial response to conventional therapy and have been undergoing treatment for less than 18 months. The trial is expected to enroll approximately 240 evaluable patients, half on the experimental arm and half on the control arm. Patients on the experimental arm will receive STR at a dose of 750 mCi/m2 plus the chemotherapy drug melphalan at 200 mg/m2, followed by autologous stem cell transplantation. Patients on the control arm will receive melphalan only, followed by transplantation. Patients on both study arms will be evaluated for response to treatment six months after transplantation, using an immunofixation assay to detect myeloma protein in patient samples. Analysis of patient samples will be conducted at a central laboratory, and blinded results will be reviewed by an independent panel of experts. The study's primary endpoint is complete response, as determined by the complete disappearance of myeloma protein at six months post-transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

1.To determine the efficacy of STR (166Ho-DOTMP). The primary endpoint of this study is to compare the CR rate at 6 months post-transplant (in the absence of further therapy) in subjects with primary refractory multiple myeloma after treatment with 750 mCi/m2 166Ho-DOTMP plus 200 mg/m2 melphalan followed by autologous PBSCT to treatment with 200 mg/m2 melphalan alone followed by autologous PBSCT.

SECONDARY OBJECTIVES:

1. To compare the treatment groups with respect to survival and progression-free survival.
2. To compare treatment groups with respect to overall response rate (CR+VGPR+PR), best response within 6 months, and duration of response.
3. To compare the safety profile of the treatment groups.
4. To assess the biodistribution and estimated radiation absorbed dose to kidney in the first 20 subjects.

METHODOLOGY: Informed consent for participation in the study will be obtained, eligibility determined, and the subject registered. All subjects will receive a tracer dose of 30 mCi 166Ho-DOTMP to determine skeletal uptake and biodistribution of 166Ho-DOTMP therapy. Subjects may receive a therapy dose only if 1) the tracer dose shows no aberrant distribution, and 2) if the skeletal residence time is at least 5.8 hours (equivalent to F x Te > 4 hr). Subjects with adequate skeletal uptake and no aberrant distribution will be stratified based on the length of time since first induction therapy, and on response to prior therapy, and will undergo randomization to determine whether they will receive 166Ho DOTMP plus melphalan (Arm A) or melphalan alone (Arm B) as the conditioning regimen prior to autologous PBSCT.

Subjects randomized to Arm A will be treated with 750 mCi/m2 166Ho DOTMP intravenously 4 to 12 days after the tracer dose, with a total dosage not to exceed 1500 mCi. Five to 9 days after the 166Ho-DOTMP therapy dose, subjects will receive 200 mg/m2 melphalan IV.

Subjects randomized to Arm B will receive 200 mg/m2 melphalan at least 10 days and no more than 3 weeks after the tracer dose.

For all patients, cryopreserved hematopoietic stem cells will be infused 24 to 48 hours after melphalan. Subjects will be followed for safety assessments for 10 years or until death. Efficacy will be evaluated for up to 3 years in responding subjects, and disease relapse or progression and survival will be documented until Year 10.

An analysis to estimate radiation dose to the kidney will be performed in the first 20 patients. Additionally, after 6 months of follow-up have been completed on the first 20 subjects in each arm, an analysis of the CR rate will be conducted to rule out lack of efficacy of 166Ho-DOTMP. A planned interim analysis to determine the efficacy of the treatment will be performed when 60 patients on each arm have completed 6 months of follow-up. Enrollment on trial will continue while these interim analyses are performed.

NUMBER OF SUBJECTS: Two hundred and forty subjects who meet the eligibility criteria and receive study treatment will be followed on this protocol.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all of the following criteria to be eligible for the study. These will be evaluated within four weeks prior to enrollment.

* Subject must have primary refractory multiple myeloma defined as having failed to achieve an objective response (CR or PR using EBMT/IBMTR/ABMTR criteria) to any therapy since the initiation of induction therapy. At least one previous therapy must be a qualifying therapy that includes high dose pulsed steroids.
* There must be < 18 months from the beginning of induction therapy to time of enrollment on study.
* Subject must meet institutional guidelines for autologous PBSCT.
* Subject must have a minimum of 2 x 106 unmanipulated CD34+ cells/kg cryopreserved and available for transplant.
* Age 18 and 70 years.
* Adequate pulmonary function defined by FEV1, FVC and DLCO > or = 50% of predicted.
* Adequate cardiac function, defined as left ventricular ejection fraction (LVEF) of > or = 45%, with no evidence of cardiac amyloidosis.
* Adequate liver function, defined as serum total bilirubin < or = 2x institutional laboratory upper limit of normal and ALT/SGPT < or = 3x institutional laboratory upper limit of normal.
* Adequate renal function, defined as 24 hour measured creatinine clearance of > or = 50 mL/min/1.73 m2 BSA and serum creatinine < or = 1.8 mg/dL.
* ECOG performance score (PS) of 0, 1, or 2.
* Women of childbearing potential must have a negative pregnancy test (serum or urine beta HCG) and be using appropriate birth control methods.
* Ability to understand the study and provide informed consent.

Exclusion Criteria:

A subject meeting any of the following criteria is not eligible for participation in the study:

* Non-secretory multiple myeloma.
* Asymptomatic MGUS, smoldering multiple myeloma, or indolent multiple myeloma.
* Solitary bone or extramedullary plasmacytoma.
* Waldenstrom's macroglobulinemia (IgM myeloma).
* Evidence of disease progression (such as new bone lesions) in the setting of a greater than 50% reduction in M-protein.
* Absence of previous therapy with pulsed corticosteroids for multiple myeloma.
* Previous high-dose therapy with stem cell or bone marrow transplant, including autologous, allogeneic, and reduced-intensity or non-myeloablative allogeneic transplants.
* Life expectancy severely limited by concomitant illness (less than 6 months).
* Evidence of symptomatic spinal cord compression or pathological fracture within 3 months.
* Cumulative external beam radiation to > 20% of marrow volume or > 40 Gy to any single region of the spinal cord.
* Prior radiation to the bladder or kidney, defined as radiation portals that directly include any volume of either kidney or the bladder.
* Uncontrolled arrhythmia or symptomatic cardiac disease.
* Clinical evidence of amyloidosis involving the heart, lungs, liver, kidney, autonomic nervous system, or GI tract.
* History of hemorrhagic cystitis.
* Current microscopic or gross hematuria in the absence of vaginal bleeding.
* Obstructive uropathy.
* Inability to have bladder catheter placed.
* Evidence of HIV-seropositivity.
* Recent history of alcohol or drug abuse.
* History of non-compliance in other studies.
* Use of bisphosphonates within 14 days preceding enrollment.
* Use of any other therapy for multiple myeloma (including standard, induction, investigational, and alternative therapies) within 4 weeks prior to enrollment.
* Experimental therapies for any other conditions in the four weeks prior to enrollment.
* Pregnant or lactating women.
* Known allergy to vitamin C or bisphosphonates.
* Other prior malignancy except for: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or any other cancer from which the subject has been disease-free for 5 years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2004-03

CONTACTS AND LOCATIONS:
Locations (21):
- United States (20):
  - University of Alabama, Birmingham, Alabama
  - Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - University of Miami, Miami, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Wayne State University, Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Giralt S, Bensinger W, Goodman M, Podoloff D, Eary J, Wendt R, Alexanian R, Weber D, Maloney D, Holmberg L, Rajandran J, Breitz H, Ghalie R, Champlin R. 166Ho-DOTMP plus melphalan followed by peripheral blood stem cell transplantation in patients with multiple myeloma: results of two phase 1/2 trials. Blood. 2003 Oct 1;102(7):2684-91. doi: 10.1182/blood-2002-10-3250. Epub 2003 May 1. PMID 12730103